CLINICAL TRIAL: NCT00743678
Title: A Phase II Study of Neoadjuvant FOLFOX6 Plus Cetuximab in Patients With Colorectal Cancer and Unresectable Liver Metastasis
Brief Title: Neoadjuvant FOLFOX6 + Cetuximab in Patients With Colorectal Cancer and Unresectable Liver Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Suk Park, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-04-018
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer; Unresectable Liver Metastasis
Keywords: Colorectal Cancer; Unresectable liver metastasis; FOLFOX6; Cetuximab; Neoadjuvant therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NEO (Experimental): NEO : Neoadjuvant therapy with FOLFOX6 plus cetuximab
  Interventions: Drug: FOLFOX6/cetuximab

INTERVENTIONS:
Drug: FOLFOX6/cetuximab — Neoadjuvant FOLFOX6/cetuximab

SUMMARY:
An innovative therapeutic strategy to increase the complete resection rate is of utmost importance in order to enhance survival in colorectal cancer patients with unresectable liver-only metastasis. Therefore, the investigators propose a prospective study of neoadjuvant chemotherapy using FOLFOX6 plus cetuximab to convert initially unresectable liver metastasis to potentially resectable disease.

DETAILED DESCRIPTION:
We will include the patients with unresectable liver-only metastatic disease independent of EGFR status. The results of this study will show the resection rate with neoadjuvant treatment in patients with colorectal cancer with liver-only metastasis.

Restaging including CT after #3, #6, #9, and #12 cycles of FOLFOX + Cetuximab

If any time, patients have PD, Off-study SD, Continue study treatment until resectable, up to #12 cycles, PD, or toxicities PR or more, If resectable, go to surgery : resection of liver metastasis and primary tumor, if present If unresectable, continue until resectable, up to #12 cycles, PD, or toxicities

Overall, a total of 12 cycles of treatment including neoadjuvant therapy will be given either before, after or without surgery.

CT scans will be performed every 3 cycles during the first 12 cycles (6 months). After that, CT scans will be performed every 2 months for another 6 months, then every 3 months for 6 months, then once a year or earlier if a PD is probable.

AEs will be evaluated once every cycle and during the CT evaluation visit.. Patients that can only undergo R1 resection or are unable to get surgery at all, will be evaluated regularly until PD.

Radiofrequency ablation (RFA) may be allowed as a palliative local therapy in patients that are suitable for it. RFA is not considered equal to a resection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal cancer with metastatic lesion(s) in the liver that is (are) unresectable
* Age ≥ 18
* ECOG performance 0 - 1
* Adequate organ function ((hepatic transaminases ≤ 5x upper limit of normal, bilirubin < 2.0 x upper limit of normal, and creatinine ≤ 1.5x upper limit of normal, platelet > 100,000/ul, absolute neutrophil count ≥ 1,500/ul)
* At least one measurable lesion by RECIST criteria
* Written informed consent

Exclusion Criteria:

* Resectable liver metastasis
* Extrahepatic metastases, regardless of their resectability
* Chronic active hepatitis or cirrhosis
* Prior therapy for metastatic disease
* Pregnant or lactating women
* Uncontrolled medical illnesses including medically uncontrolled infection, uncontrolled hypertension, unstable angina, symptomatic congestive heart failure, myocardial infarction within 6 months
* Previous adjuvant FOLFOX chemotherapy
* Prior adjuvant chemotherapy, if administered within 6 months before study entry
* Known hypersensitivity reaction to any of the components of study treatment
* Prior agents directed against EGFR
* Prior allergic reaction (known sensitivity) to chimerized or murine monoclonal antibody therapy
* Known alcohol or drug abuse
* Participation in another clinical study within the 30 days before registration
* Peripheral neuropathy > grade 1
* Other previous malignancy with exception of a history of a previous curatively treated basal cell carcinoma of the skin of pre-invasive carcinoma of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-06; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To evaluate overall R0 resection rates following neoadjuvant FOLFOX6 plus cetuximab in patients with colorectal cancer and unresectable liver-only metastasis | 18 months

SECONDARY OUTCOMES:
Response rate (according to RECIST) | 24 months
Progression-free survival time | 24 months
Overall survival timeToxicity profile (according to NCI CTCAE v3) | 24 months
Correlative analyses between pretreatment EGFR, KRAS mutation and response rate/survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Young Suk Park, M.D.,Ph.D., Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea